CLINICAL TRIAL: NCT04251390
Title: Initial Outcomes of Robotic Lower Extremity Exoskeleton Use by a Non-ambulatory Child With Cerebral Palsy: A Case Study
Brief Title: Initial Outcomes of Robotic Lower Extremity Exoskeleton Use by a Non-ambulatory Child With CP
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Elizabeth Condliffe, PhD MD, Assistant Clinical Professor, University of Calgary
Other Study IDs: REB19-1484
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy
Keywords: exoskeleton device
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- trexo Home intervention: Participants family is renting a trexo Home from trexo. The decision to use the device was separate from this research, and the decision to do research on its use was secondary. The proposed procedures may be modified to adapt to the child and family's interest and needs. Participant will use the trexo Home in their home, school, and community.
  Interventions: Device: trexo Home

INTERVENTIONS:
Device: trexo Home — 12 week intervention, with weekly contact/assessments of the affects of using the trexo Home.

SUMMARY:
There are very few evidence-based interventions for children with cerebral palsy who cannot walk. The Trexo-Home is a device that is newly available for rent by families, but its impact is unknown. By tracking and recording various outcome measures throughout this project, the investigators hope to inform future larger scale controlled studies.

DETAILED DESCRIPTION:
Design: This is a prospective case study to understand how a walking-aid device (Trexo-Home) that has been rented by a family, may impact a child with cerebral palsy (CP) who cannot walk. The decision to use the device was separate from this research, and the decision to do research on it's use was secondary, making it an observational study. The proposed procedures below may be modified to adapt to the child and family's interest and needs.

Background and Rationale: Evidence suggests that positive health outcomes are associated with reducing sedentary behaviour and sitting time. For individuals with significant motor impairments, spending the majority of their days sitting in a wheelchair is often a reality, potentially leading to secondary preventable chronic diseases such as type 2 diabetes, cardiovascular disease, and some cancers. Many children with CP have mobility limitations, and approximately 30% are non-ambulatory or require assistive devices. Currently, there are very few treatments available for non-ambulatory children with CP, and treatments may be invasive or have undesirable side effects. Tréxō Robotics (Trexo) aims to bridge the gap in treatments available for non-ambulatory children. Trexo offers a robotic exoskeleton that enables children to walk using a gait trainer with an external power source with the safety of a walker. This revolutionary technology is new to the world of pediatric rehabilitation, and Trexo Home provides the advantage of versatility to use the device at home or in the community on a daily basis. This means children who would otherwise spend most of their day sitting in a wheelchair can now stand and walk on a daily basis using this device in a familiar setting. Presently, the impacts of its use are unknown, however similar exoskeletons used with adults with spinal cord injury (SCI) show promising health benefits beyond enjoyment of walking again, such as improvements in spasticity and regularity of bowel movements.

This case study will involve one 7 year old child with CP who is functionally non-ambulatory. This child's family holds an agreement to lease the Trexo Home for a period of 6 months. Through the exploratory nature and prospective design of this case study, the investigators will gather critical data for informing future larger scale, controlled studies. With limited pediatric data related to the use of robotic assisted movement, this information could potentially add to or alter current interventions recommended for children with significant motor impairments.

Objective: The objective of this case study is to thoroughly assess the impact of Trexo Home use in one 7 year old child with CP (Gross Motor Function Classification System level IV).

i) Does using a robotic exoskeleton meet the family's primary goal - facilitating their child's experience of joy? ii) What is the family's experience around feasibility and the child's tolerability of using the Trexo at home or in the community? iii) What are the initial physiologic outcomes following twelve weeks of Trexo use?

Methods: Implementation of this project will occur over 16 weeks, with a baseline period of 4 weeks , an intervention period of 12 weeks. Throughout the project the investigators will have weekly contact with the participant's family. This frequency was selected in discussion with the family.

Joy will be evaluated using a Smiley Face Likert Scale, completed separately by the child and the parents on a weekly basis.

Feasibility and Tolerability will be quantified by number of minutes of Trexo Home use and number of steps taken per day. Reasons for skipping or abbreviating a therapeutic session will be recorded.

Physiologic outcomes evaluate key symptoms of cerebral palsy and secondary complications.

Spasticity will be assessed every second week using clinical measures (modified Tardieu and modified Ashworth Scale) and quantitative measures (the Portable Spasticity Assessment Device which differentiates reflexive and intrinsic stiffness).

Range of motion (ROM) at the hip and knee joint bilaterally will be measured via standardized goniometry, and will be done every second week, on alternate weeks from the spasticity assessment.

The child's sitting balance will be assessed monthly using the Early Clinical Assessment of Balance Version 2.

Bowel movement frequency and any related medication use will be tracked with daily diaries. This area has significant potential to enhance the quality of life of an individual, and adults with a spinal cord injury using exoskeleton have noted benefits.

Videos of the balance assessment and of free movement will occur in phase 1 and every month during phase 2, the intervention period. Video of the child using the Trexo device will be taken every two weeks in phase 2.

ELIGIBILITY:
Inclusion Criteria:

* This case study will involve one 7 year old child with cerebral palsy who is functionally non-ambulatory. This is a prospective case study to understand how a walking-aid device (trexo Home) that has been rented by a family, may impact a child with cerebral palsy who cannot walk. The decision to use the trexo exoskeleton device was separate from this research, and the decision to do research on its use was secondary.

Exclusion Criteria:

* N/A

Ages: 7 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: GMFCS IV
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Frequency of bowel movements | Daily for 12 weeks
  Daily diary describing quantity and quality of bowel movements
modified Ashworth Scale and modified Tardieu | every 1-2 weeks for 12 weeks
  Muscle spasticity measured in lower extremities
Range of motion of lower extremities | every 1-2 weeks over 12 weeks
  Standardized goniometry to measure range of ankle, knee and hip joints

SECONDARY OUTCOMES:
Early Clinical Assessment of Balance version 2 | every 1-2 weeks over 12 weeks
  Measurement tool for postural balance and head control
Parent and caregiver anecdotal reports | Weekly over 12 weeks
  To describe feasibility and tolerability of using the trexo at home or in the community
Smiley face likert scale for Joy | Daily when using the device over 12 weeks
  A scale to quantify the participant's experience of joy while using the device
Portable Spasticity Assessment Device | every 1-2 weeks over 12 weeks
  A device and software system used to measure muscle spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Condliffe, PhD, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided